CLINICAL TRIAL: NCT00274352
Title: A Double-Blind, Randomized, Placebo-Controlled Study of Adalimumab in the Treatment of Cutaneous Sarcoidosis
Brief Title: A Study of Adalimumab to Treat Sarcoidosis of the Skin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pariser, Robert J., M.D. (Other)
Collaborators: Abbott (Industry); Virginia Clinical Research, Inc. (Other)
Responsible Party: Principal Investigator, Robert J. Pariser, MD, Investigator, Virginia Clinical Research, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM05-006
Record Dates: First submitted 2006-01-06; First posted 2006-01-10 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Sarcoidosis
Keywords: sarcoidosis; adalimumab; skin diseases
MeSH Terms: conditions — Sarcoidosis; Skin Diseases | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: adalimumab — Adalimumab 40 mg administered subcutaneously once weekly or placebo injection administered once weekly for 12 weeks, followed by open-label adalimumab 40 mg administered subcutaneously weekly for an additional 12 weeks.

SUMMARY:
The purpose of this study is to determine if adalimumab is an effective for the skin manifestations of sarcoidosis.

DETAILED DESCRIPTION:
The cutaneous lesions of sarcoidosis are often disfiguring and can produce functional impairment. They tend to be hard to treat with most topical therapies and often require systemic medications which carry the risk of significant side effects. Often such treatments are withheld unless there is a need to use them for visceral involvement. There is thus an unmet need for safe and effective treatments for these patients. In addition there is essentially no controlled trial data for any treatments for cutaneous sarcoidosis. This study is intended to determine if adalimumab might offer a viable therapeutic option for this condition by comparing the response of cutaneous sarcoid lesions to this drug as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age.
2. Subject must have moderate to severe cutaneous sarcoidosis with chronic indurated lesions (papules, nodules, and/or plaques), which histopathologically show non-caseating granulomas with negative special stains for microorganisms (AFB and PAS or GMS). Accepted clinical variants include, but are not necessarily limited to the following:

   * lupus pernio
   * nodular
   * subcutaneous
   * annular
   * angiolupoid
   * plaque
   * papular
   * lichenoid
   * psoriasiform
3. For purposes of this study "moderate to severe cutaneous sarcoidosis" is defined as the presence of sarcoidal skin lesions with any of the following features:

   * At least 5 easily visible facial lesions, or
   * Disease which involves > 3% BSA, or
   * Disease which confers functional impairment (e.g. nasal or visual field obstruction), or
   * Disease which confers significant symptoms of itching and/or pain.
4. If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or is using one of the following methods of birth control for the duration of the study and 90 days after study completion:

   * condoms, sponge, foams, jellies, diaphragm, or intrauterine device
   * contraceptives (oral or parenteral) for three months prior to study drug administration
   * a vasectomized sole partner
5. Females of childbearing potential must have a negative serum pregnancy test at screening visit.
6. Subject must have no history of nor evidence of tuberculosis, either active or previously treated. This determination will be based on a negative PPD skin test and negative chest radiograph at screening, negative history of previous tuberculosis, and negative history of previous exposure to tuberculosis.
7. Subject must be willing and able to give informed consent and to comply with the requirements of the protocol.
8. Subject must be willing and able to self-administer SC injections or to have a qualified person available to administer SC injections.
9. The following criteria for concomitant treatments of sarcoidosis must be met:

   * Topical therapies (corticosteroids) must be discontinued at least 2 weeks prior to baseline visit.
   * Intralesional therapies (corticosteroids) must be discontinued at least 4 weeks prior to baseline visit.
   * Systemic therapies (MTX, antimalarials, prednisone, immunosuppressants, thalidomide, tetracycline derivatives) must be discontinued at least 4 weeks prior to baseline visit.

OR if a subject is on such topical or oral medications, the dose has been stable for these same time intervals and is likely to remain stable for the duration of the study. Patients whose non-cutaneous disease is being managed by other physicians will continue to have their care directed by these physicians. The managing physicians will be kept informed of the patients' status, consistent with study blinding. If the patient's dose of a concomitant systemic therapy for non-cutaneous sarcoidosis must change by more than 20% of the dose at study entry due to a change in medical condition during the double-blind phase, the subject will be discontinued from the study. During the open-label phase the need for a greater than 20% increase in dose of concomitant treatment for non-cutaneous sarcoidosis will be viewed as treatment failure and the patient will be discontinued from the study. Reduction of the dose of such treatment of any magnitude will not result in discontinuance. Continued use of intralesional therapies is not permitted. Inhaled corticosteroids for a stable medical condition are allowed.

Exclusion Criteria:

1. Evidence of other active skin diseases or skin infections during screening that may interfere with evaluation of sarcoidosis.
2. Subject has a known sensitivity to any component of the study medication. (See Table 4.)
3. Subject has an active infection requiring systemic antibiotics at time of screening.
4. Subject has a history of malignancy or lymphoproliferative disease within the past 5 years, excluding successfully treated non-melanoma epithelial skin cancer and/or localized carcinoma in situ of the cervix.
5. Subject has a history of congestive heart failure.
6. Subject has a poorly controlled medical condition including, but not limited to, unstable cardiovascular disease, poorly controlled diabetes, recent stroke, history of recurrent infections, or any other condition for which, in the opinion of the investigator, participation in the study would place the subject at risk.
7. Subject has a history of demyelinating CNS disease.
8. Subject has a history of listeriosis, treated or untreated tuberculosis, exposure to individuals with tuberculosis, persistent or active infections requiring hospitalization or treatment with IV antibiotics, IV antiretrovirals, or IV antifungals within 30 days of baseline, OR oral antibiotics, antivirals, or antifungals for purpose of treating infection, within 14 days of baseline.
9. Subject is currently using or plans to use antiretroviral therapy at any time prior to or during study.
10. Previous use of anti-TNF agent(s).
11. Receipt of any other investigational product within 30 days prior to the first dose of investigational product.
12. Subject is known to have immune deficiency or is immunocompromised.
13. Female subjects who are pregnant, breast feeding, or are considering becoming pregnant during the study or within 150 days of the last dose of study medication.
14. Subject has a history of clinically significant drug or alcohol abuse in the last year.
15. Subject is considered by the investigator, for any reason, to be an unsuitable candidate for study participation.
16. Clinically significant ECG abnormalities at screening visit.
17. Hgb < 8.5 g/dL in females and < 9.0 in males.
18. WBC count < 3000/mm2
19. AST or ALT > 2.0 times the upper limit of normal for the age range, confirmed by a repeat measure.
20. Bilirubin > 3mg/dL
21. Creatinine > 1.6 mg/dL in women, and > 1.8 mg/dL in men.
22. Subject plans to receive any live vaccines during the study.
23. Subject has a variant of sarcoidosis that is not amenable to study evaluation, in the absence of chronic indurated lesions, such as:

    * Acute, "benign" sarcoid associated with erythema nodosum
    * Acute iritis
    * Ichthyosiform sarcoidosis
    * Hypo- or hyperpigmented macular sarcoidosis
    * Ulcerative sarcoidosis
    * Erythroderma
    * Alopecia

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who are Responders, achieving at least Moderate Improvement on the Physician's Global Assessment, after 12 weeks of treatment during Period A (double-blind phase). | at completion of double-blind phase (12 weeks)

SECONDARY OUTCOMES:
Proportion of subjects achieving a PGA (Physician's Global Assessment) of Clear or Marked Improvement after 12 weeks of treatment during Period A. | at completion of double-blind phase (12 weeks)
Proportion of subjects achieving at least a PGA of Mild Improvement after 12 weeks of treatment during Period A. | at completion of double-blind phase (12 weeks)
Change in the patient's Quality of Life score relative to baseline after 12 weeks of treatment during Period A. | at completion of double-blind phase (12 weeks)
Change in the Patient's Global Assessment relative to baseline after 12 weeks of treatment during Period A. | at completion of double-blind phase (12 weeks)
Proportion of subjects with a 12% or greater improvement (minimum of 200mL change) in FVC and/or FEV1 after 12 weeks of treatment during Period A. (This is the minimum change thought to be clinically significant per American Thoracic Society Statement | at completion of double-blind phase (12 weeks)
Proportion of subjects with improvement in pulmonary diffusing capacity after 12 weeks of treatment during Period A. | at completion of double-blind phase (12 weeks)
Proportion of subjects with observed improvement on chest radiograph after 12 weeks of treatment during Period A. | at completion of double-blind phase (12 weeks)
(Sub group analysis of all subjects by CXR stage at study entry will be performed for all respiratory variables) | at completion of double-blind phase (12 weeks)
Change target lesion dimensions and estimated thickness. | at completion of double-blind phase (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Pariser, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Virginia Clinical Research, Inc., Norfolk, Virginia, United States